CLINICAL TRIAL: NCT07019818
Title: Esmolol Versus Sufentanil on the Quality of Recovery After Laparoscopic Cholecystectomy During Anaesthesia With Orotracheal Intubation on an Outpatient Basis
Brief Title: Esmolol Versus Sufentanil on the Quality of Post-cholecystectomy Recovery Laparoscopic Anaesthesia With Orotracheal Intubation on an Outpatient Basis
Acronym: ESA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 87RI_24_0041 - ESA; 2024-520282-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-13; First posted 2025-06-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Laparoscopic Cholecystectomy Surgery
MeSH Terms: interventions — esmolol; Sufentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (experimental arm) (Experimental): Esmolol 1 à 1,5 mg/kg at induction
  Interventions: Drug: Esmolol Hcl 10Mg/Ml Inj
- Group 2 (comparator arm) (Active Comparator): Sufentanil 0,1 à 0,3 μg /kg at induction.
  Interventions: Drug: Sufentanil 5 mcg

INTERVENTIONS:
Drug: Esmolol Hcl 10Mg/Ml Inj — Esmolol is an injectable cardioselective beta-blocker, preferentially inhibiting beta-1 adrenergic receptors, while avoiding an increase in peripheral vascular resistance.
  Arms: Group 1 (experimental arm)
Drug: Sufentanil 5 mcg — Sufentanil is a synthetic opioid with the pharmacological properties of a µ-receptor agonist.
  Arms: Group 2 (comparator arm)

SUMMARY:
There are 120,000 outpatient laparoscopic cholecystectomies with orotracheal intubation per year in France.

Sufentanil is the most commonly used morphine during surgery in France, but morphines have harmful effects when administered for surgery. As with other morphine-based analgesics (painkillers), sufentanil can be associated with nausea and vomiting, confusion, itching and addiction.

There is an approach to anaesthesia which aims to eliminate the use of morphine in order to avoid its side effects, but there is a lack of clinical trials and benchmarks to provide proof of this.

Esmolol is a cardioselective beta-blocker (a substance that acts only on the heart) which also has marketing authorisation for all types of surgery, the most frequent side effects of which are hypotension and bronchospasm.

These two drugs have different therapeutic properties for a common objective under general anaesthesia, namely the stability of vital parameters (such as pulse, blood pressure, blood oxygenation, etc.) during surgery.

Esmolol disappears very quickly from the body, which could give it an interesting place in outpatient management.

The hypothesis tested in this study is that the use of Esmolol is an effective alternative to Sufentanil during general anaesthesia for laparoscopic cholecystectomy with orotracheal intubation on the quality of post-operative recovery and pain.

The aim of this study is to evaluate whether the use of Esmolol is equivalent to the use of Sufentanil in terms of patient comfort, assessed in terms of quality of recovery, after general anaesthesia with orotracheal intubation for laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The study will recruit 120 patients over a period of 18 months. Each patient will participate for two days.

The study is multicentre, which means that patients from several hospitals will be able to take part. Two hospitals will be taking part: Brive La Gaillarde Hospital and Limoges University Hospital.

The aim of this equivalence study is to compare Esmolol with Sufentanil. If you agree, and after the study doctor has checked the inclusion criteria and provided you with information, you will sign a consent form.

In this study, we are going to compare two different anaesthetic treatments:

* Group 1: use of Esmolol
* Group 2: use of Sufentanil Regardless of the group, as part of this study, you will receive one day's follow-up which will consist of a single visit by telephone by a member of the team, during which you will be asked to complete a short questionnaire on the quality of recovery the day after your surgery and you will also be asked about your consumption of painkillers at home.

This research is open to all adult patients, in good health or suffering from a mild or severe non-life-threatening condition, scheduled for laparoscopic cholecystectomy as an outpatient, under general anaesthetic with orotracheal intubation (which consists of placing a tube in the trachea through the glottic orifice, with the upper end emerging through the mouth, a routine procedure in the operating theatre).

Unfortunately, however, you cannot take part if you are taking beta-blockers or if you have any contraindications to taking beta-blockers; or if you have uncontrolled hypertension or abnormal vital parameters (pulse, blood pressure); or if you are expected to have difficulty intubating during the anaesthetic consultation, or if you are severely obese. You may also not take part if you are pregnant or breastfeeding, or if you are hypersensitive to the active substance or to any of the excipients of sufentanil and esmolol, or if you are under guardianship or deprived of your liberty.

You will receive a medical examination during your anaesthetic consultation. Participating patients must be affiliated to a social security scheme.

If you take part in this research, there will be three visits:

* An inclusion visit, which will take place during your anaesthetic consultation, where the investigating doctor will check the eligibility criteria and collect your written consent to take part. Data will be collected: age, sex, comorbidities (obstructive ventilatory disorders (asthma/BPCO) and opiate addiction), clinical characteristics such as weight, height, BMI, ASA score, heart rate, blood pressure.
* A 2nd visit on the day of your surgery, when the investigating doctor will double-check certain eligibility criteria (use of beta-blockers, cancelled cholecystectomy, pregnancy) and then draw lots by computer to decide which group you will be in (group 1: esmolol or group 2: sufentanil), with vital parameters recorded.
* A 3rd and final visit the day after your surgery, during which a quality of recovery questionnaire (15 questions) will be completed over the telephone by a member of the team, as well as an assessment of your consumption of painkillers at home.

You will not know which group you are in, so as not to influence your answers to the quality of recovery questionnaire carried out by telephone the day after your surgery; nor will the person who contacts you to ask you the questions. However, your doctor will know which group you are in.

Your doctor must provide you with all the necessary explanations concerning this research. If you wish to withdraw at any time, for whatever reason, you will continue to benefit from medical monitoring and this will in no way affect your future surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* ASA I to III
* Scheduled outpatient cholecystectomy
* General anesthesia with orotracheal intubation
* Patient with signed consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patients on beta-blockers
* Uncontrolled hypertension
* Contraindication to beta-blockers
* Hypersensitivity to the active substance or to one of the excipients of sufentanil and esmolol
* Pre-existing hemodynamic abnormality
* Intubation planned to be difficult during the anaesthesia consultation
* Severe obesity (BMI > 35 kg/m2)
* Pregnant or breast-feeding women
* Patients deprived of liberty
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-02 (Estimated); Primary Completion 2028-01-04 (Estimated); Study Completion 2028-01-05 (Estimated)

PRIMARY OUTCOMES:
To Describe the difference in quality of recovery using the questionnaire | 2 days
  To estimate the difference in the quality of recovery score (fQoR-15) at D1 between the two randomisation groups (Esmolol versus Sufentanil), as well as its 95% confidence interval.

IPD SHARING:
Plan to Share IPD: No